CLINICAL TRIAL: NCT03009357
Title: Clinical Application of Continuous Monitoring Data for the Pulse Rate, Exercise, and Calorie Intake by Wearable Activity Trackers in the Patients With Thyrotoxicosis
Brief Title: Clinical Application of Pulse Rate-monitoring Activity Trackers in Thyrotoxicosis
Acronym: AT-thyro
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae Hoon Moon, Assistant professor, Seoul National University Bundang Hospital
Other Study IDs: B-1609/363-004
Record Dates: First submitted 2016-12-29; First posted 2017-01-04 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Thyrotoxicosis; Graves Disease; Thyroiditis
Keywords: wearable activity tracker; thyrotoxicosis
MeSH Terms: conditions — Thyrotoxicosis; Graves Disease; Thyroiditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- thyrotoxicosis: patients with newly detected or recurrent thyrotoxicosis
- control: euthyroid, healthy adults

SUMMARY:
The study is a single-center prospective cohort study of clinical application of continuously monitored data by wearable activity trackers in the patients with thyrotoxicosis. The purpose of the study is to evaluate the association between parameters of pulse rate, activity, and sleep from wearable activity trackers and the thyrotoxic status along with the treatment.

DETAILED DESCRIPTION:
Activity trackers to be used: Fitbit Charge HR (TM)

Data which ware provided by Fitbit app (TM) will be analyzed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing newly developed or recurrent thyrotoxicosis who are treated and followed-up in Seoul National University Bundang Hospital
* Patients who can use wearable activity trackers and smartphone applications
* In case of Graves' disease, patients who will treated by anti-thyroid drugs

Exclusion Criteria:

* Patients who have thyrotoxic periodic paralysis
* In case of Graves' disease, patients who will treated by radioactive iodine therapy or thyroidectomy
* Patients who have thyrotoxicosis due to toxic nodular disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults (20 to 60 years) undergoing newly developed or recurrent thyrotoxicosis who can use wearable activity trackers and smartphone applications
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Association between parameters of pulse rate, activity, and sleep from wearable activity trackers and the thyrotoxic status | continuous monitoring through the study period (average 3 months)

SECONDARY OUTCOMES:
Association between user-generated dietary parameters on mobile applications and the thyrotoxic status | continuous monitoring through the study period (average 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hoon Moon, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JE, Lee DH, Oh TJ, Kim KM, Choi SH, Lim S, Park YJ, Park DJ, Jang HC, Moon JH. Clinical Feasibility of Monitoring Resting Heart Rate Using a Wearable Activity Tracker in Patients With Thyrotoxicosis: Prospective Longitudinal Observational Study. JMIR Mhealth Uhealth. 2018 Jul 13;6(7):e159. doi: 10.2196/mhealth.9884. PMID 30006328
- [Derived] Lee JE, Lee DH, Oh TJ, Kim KM, Choi SH, Lim S, Park YJ, Park DJ, Jang HC, Moon JH. Clinical Feasibility of Continuously Monitored Data for Heart Rate, Physical Activity, and Sleeping by Wearable Activity Trackers in Patients with Thyrotoxicosis: Protocol for a Prospective Longitudinal Observational Study. JMIR Res Protoc. 2018 Feb 21;7(2):e49. doi: 10.2196/resprot.8119. PMID 29467121